CLINICAL TRIAL: NCT03178240
Title: Randomized Trial of a Photoaging Mirroring Intervention for Skin Cancer Prevention in Secondary Schools in Brazil - Study Protocol
Brief Title: Sunface Mirroring RCT in Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Titus J. Brinker, Titus J. Brinker, MD, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SunfaceMirrorBrazil
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 45 minutes seminar on skin cancer prevention and UV-protection in general.
  Interventions: Behavioral: photoaging mirroring intervention
- Control (No Intervention): The control croup takes part in the survey but does not receive an intervention.

INTERVENTIONS:
Behavioral: photoaging mirroring intervention — selfies of the students are photoaged showing them the consequences of their UV protection behavior on their own face
  Arms: Intervention

SUMMARY:
Randomized trial looking at the effects of a behavioral photoaging software intervention on sunscreen use in the city of Itauna, Brazil.

ELIGIBILITY:
Inclusion Criteria:

Visiting a secondary school in Brazil.

Exclusion Criteria:

Not visiting a secondary school in Brazil.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in prevalence of daily sunscreen use at six months | 6 months
  The difference between daily sunscreen use in the past 30 days in the intervention group from baseline to six months follow-up vs. in the control group from baseline to six months follow-up.
Change in prevalence of daily sunscreen use at one months | 1 month
  The difference between daily sunscreen use in the past 30 days in the intervention group from baseline to one months follow-up vs. in the control group from baseline to one month follow-up.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brinker TJ, Faria BL, de Faria OM, Klode J, Schadendorf D, Utikal JS, Mons U, Krieghoff-Henning E, Lisboa OC, Oliveira ACC, Lino HA, Bernardes-Souza B. Effect of a Face-Aging Mobile App-Based Intervention on Skin Cancer Protection Behavior in Secondary Schools in Brazil: A Cluster-Randomized Clinical Trial. JAMA Dermatol. 2020 Jul 1;156(7):737-745. doi: 10.1001/jamadermatol.2020.0511. PMID 32374352
- [Derived] Brinker TJ, Faria BL, Gatzka M, de Faria OM, Heppt MV, Kirchberger MC, Schadendorf D, Nakamura Y, Buslaff F, Lisboa OC, Oliveira ACC, Lino HA, Bernardes-Souza B. A skin cancer prevention photoageing intervention for secondary schools in Brazil delivered by medical students: protocol for a randomised controlled trial. BMJ Open. 2018 Mar 6;8(3):e018299. doi: 10.1136/bmjopen-2017-018299. PMID 29511007